CLINICAL TRIAL: NCT03781765
Title: Stimulant vs. Non-stimulant Treatments and Reward Processing in Drug-naive Youth at SUD Risk
Acronym: MPH-ATX
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Jeffrey Newcorn, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: GCO 17-0423; 1R21DA045218-01A1 (NIH)
Record Dates: First submitted 2018-12-18; First posted 2018-12-20 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: ADHD; Attention Deficit Hyperactivity Disorder
Keywords: fMRI Study; MPH; Methylphenidate; ATX; Atomoxetine; Reward System; Substance Abuse Risk
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate; 5,10-dihydro-5-methylphenazine; Atomoxetine Hydrochloride

STUDY DESIGN:
Intervention Model Description: This is a pilot study with no control group. All youth will be treated with MPH or ATX and receive pre and post fMRI.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Methylphenidate (Active Comparator): 0.5 mg/kg for 1 week and 1 mg/kg for 2 weeks
  Interventions: Drug: Methylphenidate
- Atomoxetine (Active Comparator): 0.5 mg/kg for 1 week and 1 mg/kg for 2 weeks
  Interventions: Drug: Atomoxetine

INTERVENTIONS:
Drug: Methylphenidate — stimulant medication
  Other Names: MPH
  Arms: Methylphenidate
Drug: Atomoxetine — non-stimulant medication
  Other Names: ATX
  Arms: Atomoxetine

SUMMARY:
The study team will examine the effects of FDA approved stimulant and non-stimulant medications for ADHD, among youth with ADHD and with and without Oppositional Defiant Disorder (ODD) or Conduct Disorder (CD), on reward systems of the brain using fMRI.

DETAILED DESCRIPTION:
Longitudinal studies have shown that childhood Attention Deficit/Hyperactivity Disorder (ADHD) and child disruptive behavior disorders play an important role in the development of later Substance Use Disorders (SUD). Although available evidence suggests that abnormal reward processing is likely to mediate vulnerability for addiction, the functioning of the brain reward systems in at-risk individuals preceding the exposure to drugs remains largely unknown. Better understanding the baseline characteristics of reward processing in drug-naïve individuals at risk for later SUD is an important initial step in refining our knowledge of the neurobiological basis of addiction. Reward processing in at-risk individuals may be further influenced by exposure to first-line treatments (e.g. methylphenidate (MPH)) for ADHD that also happen to be controlled substances.

Findings from animal research have raised the possibility that stimulants such as methylphenidate (MPH) may have "sensitization" effects - which prime the brain reward system for enhanced responding to the rewarding effects of abusable substances, whereas non-stimulants such as atomoxetine (ATX) may diminish drug self-administration. However, no studies have examined the purported different effects of stimulants vs. non-stimulants on the brain reward system utilizing a targeted biomarker approach linked to an a priori model, which focuses on intermediate phenotypes. Such research could provide important knowledge regarding the biological basis of addiction vulnerability and aid in the development of preventive interventions.

This proposal will provide pilot data for the hypotheses that stimulant and non-stimulant medications have differential effects on activation in the brain reward system in High Risk (HR) youth, and that differences activation will be related to changes in measures of reward sensitivity on psychometric tests. The study team believes that this protocol is uniquely innovative in its approach to study drug-naïve children at the highest levels of risk for SUD, thus providing an opportunity to delineate differential effects of medication treatment in relation to SUD risk. This research is also significant since it will be the first neuroimaging study to assess the biological correlates of the effects of stimulants on reward sensitivity in HR children, and especially in relation to purported changes in reward processing.

ELIGIBILITY:
Inclusion Criteria:

* Pre-pubertal (e.g. Tanner stage 1 or 2)
* Age 7-12 inclusive
* Signed consent/assent
* Parent communicates sufficiently in English to provide informed consent and complete assessment instruments;
* ADHD as determined by computerized DISC (C-DISC) parent interview
* ADHD-Rating Scale-5 total score (interview with parent )
* SNAP ADHD total score (teacher) of 1.5 SD > age/sex norms
* CD or severe ODD: CD or ODD + 2 symptoms of CD on C-DISC
* SNAP ODD/CD subscale (parent and teacher) 1.5 SD > age/sex norms

Exclusion Criteria:

* Major neurological/medical illness
* History of head injury
* Fetal exposure to alcohol/drugs
* Diagnosis of major psychiatric disorder (e.g., schizophrenia, bipolar disorder, major depression, generalized anxiety, social phobia, Tourette's Disorder, PTSD, autism spectrum disorder)
* Current suicidal ideation or past history of suicide attempt
* Wechsler Abbreviated Scale of Intelligence (WASI)75 score <75
* Prior or current treatment with stimulants (prior or current treatment with non-stimulants is permitted, but participants must be off medication for 2 weeks at baseline)
* Current or past alcohol/drug use (DISC interview; urine toxicology)
* Psychological or medical condition which precludes being in the scanner (e.g., claustrophobia, morbid obesity)
* Metal in the body that cannot be removed (e.g., braces, metal plate)
* Visual disturbances that may impair task performance
* Precocious puberty (e.g. Tanner stage >2) or pregnancy

Notes:

* History of SUD in a 1st degree relative is permitted, and is expected in ~1/2 of the subjects
* Ongoing psychosocial treatment is allowed but should not be initiated during the study

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Estimated)
Dates: Start 2019-06-04 (Actual); Primary Completion 2025-09-25 (Estimated); Study Completion 2025-09-25 (Estimated)

PRIMARY OUTCOMES:
fMRI Measure | 3 Weeks
  Bold activation change within the reward system (e.g., ventral striatum, insula and orbitofrontal cortex)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Newcorn, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Iliyan Ivanov, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No